CLINICAL TRIAL: NCT00907491
Title: Use of Objective Cough Counting Device to Assess the Accuracy of Cough Detection in Healthy Adults Simulating Cough in Different Postures, Mobility and Environmental Conditions
Brief Title: Accuracy of Cough Detection in Healthy Adults
Status: Completed | Type: Observational
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Dr. Hanna Levy - Director of clinical studies, KarmelSonix Ltd
Other Study IDs: WIM-CC 01
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2009-05

CONDITIONS: Cough
Keywords: Cough; Wheeze Rate; Respiratory Function Tests
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Device: pulmonary sounds analyzer

INTERVENTIONS:
Device: pulmonary sounds analyzer — Cough counting device based on the WIM Technology

SUMMARY:
Cough is part of the defense mechanism to protect the lung from foreign particles and remove secretions from the airways. However, at times it becomes a bothersome, annoying symptom that interferes with the quality of life, sleep pattern and exercise tolerance of the patient.

People with respiratory infection, asthmatic patients and CF patients suffer from a multitude of pathologies of airways and are often inflicted with chronic cough.

Treatment of cough in these patients consists of many types of expectorants, cough suppressors, secretion modifiers, inhaled bronchodilators etc. In addition, chest physical therapy (PT) is often prescribed as part of the treatment regime.

The primary objective of the study is to evaluate the efficacy and validity of novel cough counting device based on the WIM Technology.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent
* Patients above 21 years old
* No medical history

Exclusion Criteria:

* Skin lesions precluding attachment of sensors
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults 21 years and above
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To evaluate cough detection and counting technology (ACCA) for adult people in different recording conditions | within 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel